CLINICAL TRIAL: NCT04345302
Title: Brief Motivational Therapy Versus Enhanced Usual Care for Alcohol Use Disorder in Primary Care in Chile, an Exploratory Randomised Trial
Brief Title: Brief Motivational Therapy Versus Usual Care for Alcohol Use Disorders in Primary Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nicolás Barticevic (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor-Investigator, Nicolás Barticevic, Principal Investigator, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONDECYT 11190874
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Use Disorder
Keywords: Primary care; Alcohol use disorder; Motivational interview
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: The study is a parallel-group, single-blinded, randomized clinical trial to test the superiority of a Brief Motivational Treatment over enhanced usual care. The allocation ratio is 1:1 as per a computer-generated randomisation schedule stratified by site and the baseline SDSS-DAYS score using permuted blocks of random sizes.
Who Masked: Outcomes Assessor
Masking Description: A research assistant blinded to the allocation of the participant will perform the follow-up assessments. Due to the nature of the intervention, the participants and the therapists will know in which group they are participating; however, they will be strongly instructed to not disclose their allocation at the follow-up assessments. At trial closure, a statistician blinded to allocation will conduct the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief motivational treatment (Experimental): Participants in the intervention group will receive the Brief Motivational Treatment, which is a primary care-adaptation of the Motivational Enhancement Therapy as manualized in the Project MATCH [19]. This treatment consists of four 45-minute sessions, provided by a psychologist at weeks one, two, six, and twelve. The first three sessions, occurring during the first six weeks, are more active regarding the behavioural change, while the last session functions as closure and review of the process. If a participant asks for more support, they will be able to attend up to two extra sessions before the last one.
  The main adaptations are:
  * The translation into Chilean Spanish.
  * Update of Motivational Interview concepts.
  * Companion training material that includes a demonstrative video and practical exercises.
  * An adapted personalized feedback procedure.
  * Information on additional resources available in the primary care centre and the community.
  Interventions: Behavioral: Brief motivational treatment; Behavioral: Enhanced Usual Care
- Enhanced usual care (Active Comparator): All participants will receive an educational brochure on alcohol use disorder, with self-help materials and guides on how to get additional support.
  The physicians within the PC centre will also receive information on how to diagnose alcohol use disorders, prescription guides for the medications that are available for treating these disorders in the PC centre (mainly Disulfiram and any other if available), and directions on when and where to refer clients for treatment.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Brief motivational treatment — The treatment will be delivered by general psychologists with at least three years of experience in primary care. They will receive training and then will demonstrate proficiency in a simulated client session.
  During recruitment, therapy sessions will be recorded, and ten percent of them will be reviewed using a proficiency scale. Then, a feedback report will be issued and discussed with each therapist.
  Arms: Brief motivational treatment
Behavioral: Enhanced Usual Care — During the trial, participants will continue to receive regular medical and social care at their health centre. These services may include prescriptions for mental health issues and alcohol (Disulfiram, anti-craving, anti-depressants, and other medications), social assistance, and the full spectrum of primary health care. Nevertheless, they will not receive other psychosocial interventions for alcohol use disorder in the health centre.

SUMMARY:
Harmful alcohol use is a leading cause of global disability and death. However increased detection and brief intervention capacity of more severe alcohol use disorders (AUD) has not been accompanied by increased availability of treatment services. Incorporating treatment for such disorders into primary care (PC) is of paramount importance for improving access and health outcomes. This study aims to estimate the effectiveness of a Brief Motivational Treatment (BMT) applied in primary care for treatment of these disorders.

This trial aims to test the superiority of BMT over enhanced usual care with a reasonable margin, over which the BMT could be further considered for incorporation into PC in Chile. Its pragmatic approach ultimately aims to inform policymakers about the benefit of including a brief psychosocial treatment into PC.

DETAILED DESCRIPTION:
This exploratory trial aims to estimate the effectiveness of a BMT for AUD provided in PC. The underlying question is whether Chilean PC should incorporate this treatment among its regular programs based on its effectiveness.

To answer this question, a randomised comparison between the manualized BMT and EUC will be undertaken. The main hypothesis is a superiority one:

• Participants under BMT will perform better than EUC in the reduction of alcohol consumption.

Also, there are ancillary questions that deserve special attention. The following hypotheses will help with the explanation of the results:

* Active BMT components (i.e., the working alliance and fidelity to the MI strategies) mediate the effect.
* Participant´s AUD severity mediates the effect.
* Participants under BMT will receive a higher amount of additional care (physician consultations, social worker consultations, participation in alcoholic anonymous, and others).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of alcohol use disorder according to the DSM-V (American Psychiatric Association, 2013
* Must fulfill criteria for alcohol use disorder and criteria for harmful alcohol use during the last month, i.e., five or more heavy drinking occasions in the last month (5 or more drinks in men, 4 or more in women), or an average use of 14 or more drinks a week in men, and 7 or more in women
* Also, alcohol use should be the main problem motivating participants to seek treatment.

Exclusion Criteria:

* Clients under 20 years old
* Clients in whom alcohol use is not the main problem
* Clients who leave the area or are unable for follow-up contact
* Clients with severe mental comorbidity
* Clients with severe cognitive impairment, illiteracy, or unable to follow treatment in Spanish.
* Clients who are concurrently receiving or planning to receive other psychosocial treatment for alcohol use disorder other than usual care, i.e., formal professional treatment outside of primary care. Participation in community services and Alcoholics Anonymous is permissible.
* Clients who have previously participated in the study, or whose family members are or have been participants.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in the Drinks per Drinking Day (DDD) | Baseline and six-months follow-up
  The change from baseline in the DDD during the last 90 days. The DDD will be aggregated using means.

SECONDARY OUTCOMES:
Change in the alcohol use pattern | Baseline and six-months follow-up
  The number of participants with a low-risk alcohol use pattern estimated by the number of days of consumption, of abstinence, and intoxication during the last 90 days, aggregated using the proportion of participants per group.
Abstinence days | At six-months follow-up
  The most extended period of abstinence since enrolment. The number of abstinence days of each participant will be aggregated using means.
Change in the negative consequences of alcohol use | Baseline and six-months follow-up
  The change from baseline in the negative secondary consequences of alcohol consumption will be measured using the Drinker Inventory of Consequences (DrInC-2R) questionnaire, and will be aggregated using means. The DrInC-2R has a score range from 0 to 150, with higher scores indicating higher consequences.
Change in the severity of the dependency | Baseline and six-months follow-up
  The change from baseline in the severity of the alcohol use disorder using the Substance Dependence Severity Scale. Means will be used to aggregate participants' DAYS, SEV, and WORST SEV scores for alcohol.
  The DAYS score varies on an 8-point scale ranging from 0 (symptom did not occur) to 7 (symptom occurred every day of past 30). The SEV and WORST SEV severity variables are scored on a 6-point scale ranging from 0 (absent) to 5 (extreme), with a score of '2' indicating that the diagnostic criterion has been met. Lower scales scores represent less severe dependence, and higher scale scores reflect more severe dependence.
Change in the motivation for change | Baseline and six-months follow-up
  The change from baseline in the motivational stage measured with the Stages of Change Readiness and Treatment Eagerness Scale-Drug (SOCRATES). The proportion of participants that improve their motivational stage will be used to aggregate the measurement in each group. The SOCRATES scores range within three dimensions: Recognition (7 - 35), Ambivalence (4 - 20), and Taking Steps (8 - 40), with higher scores indicating higher involvement in the dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Barticevic, MD, Principal Investigator — Adjunct Professor School of Medicine Pontificia Universidad Catolica de Chile
Locations (3):
- Chile (3):
  - CESFAM Juan Pablo II, Santiago
  - CESFAM Madre Teresa de Calcuta, Santiago
  - CESFAM San Alberto Hurtado, Santiago

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, dataset, and statistical code are available in the Open Science Foundation repository, DOI 10.17605/OSF.IO/6BA3W
Supporting Information: Study Protocol, SAP
Time Frame: From protocol registration on.
Access Criteria: Public
URL: https://doi.org/10.17605/OSF.IO/6BA3W

REFERENCES:
- [Derived] Barticevic NA, Poblete F, Zuzulich SM, Rodriguez V, Bradshaw L. Brief motivational therapy versus enhanced usual care for alcohol use disorders in primary care in Chile: study protocol for an exploratory randomized trial. Trials. 2020 Jul 31;21(1):692. doi: 10.1186/s13063-020-04589-4. PMID 32736578